CLINICAL TRIAL: NCT02417714
Title: Prospective Evaluation of Next Generation CT Reconstruction
Brief Title: Prospective Evaluation of Next Generation CT Reconstruction (NextGenIR)
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140188; 14-H-0188
Record Dates: First submitted 2015-04-15; First posted 2015-04-16 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-10-29

CONDITIONS: Healthy Subjects
Keywords: Computed Tomography; Radiation Reduction; Iterative Reconstruction; Natural History

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Body CT group: 100 subjects for a body CT
- Chest Ct Group: 115 subjects for a chest CT

SUMMARY:
Background:

- Computed Tomography (CT) is a scan that makes detailed pictures of the body. It uses radiation to do that. In 2011, about 85.3 million CT scans were done in the United States. But there is growing concern about the health effects of radiation. There are new and different ways to make CT pictures that use less radiation. Researchers want to learn whether these new methods create images that are similar to images from a traditional CT.

Objective:

- To learn if new CT imaging methods with less radiation make images that are similar to traditional ways.

Eligibility:

- Adults 18 years of age and older who are scheduled for a CT of the chest, abdomen and pelvis with contrast.

Design:

* Researchers will review participants medical records to see if they can be in this study.
* Participants may have blood drawn from an arm vein by a needle stick. The blood will be used to make sure they can be in this study and that it is safe for them to have contrast.
* During the participants CT scan appointment, one extra scan will be done using low radiation methods.
* During a CT scan, the participant lies on a table. A large x-ray machine takes pictures of the body.

DETAILED DESCRIPTION:
Computed Tomography uses ionizing radiation to make pictures of the body. Different methods of creating CT pictures have been developed that allow reductions in the amount of radiation. The purpose of this research study is to learn whether these new imaging methods using less radiation to create images are similar to the traditional and current method.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria for Body CT:

1. Clinical indication for a chest, abdomen and pelvis CT with contrast
2. Age equal to or greater than 18 years
3. Able to understand and willing to sign the Informed Consent Form

Inclusion Criteria for Chest CT:

1. Clinical indication for a CT with or without contrast that includes the chest
2. Age equal to or greater than 18 years
3. Able to understand and willing to sign the Informed Consent Form

EXCLUSION CRITERIA:

Exclusion Criteria for Body CT:

1. Pregnancy
2. Serum Cr > 1.5 mg/dL
3. Clinical CT scan with more than one contrast imaging phase (for example three phase liver)

Exclusion Criteria for Chest CT

1. Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be enrolled at the NIH Clinical Center. A total of 215 subjects will be enrolled. Subjects will be recruited from the NIH Clinical Center radiology department from subjects scheduled to have a CT scan of the chest, abdomen and pelvis with contrast.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Estimated)
Dates: Start 2014-09-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Compare with respect to 6 image quality metrics the overall image quality from a research low radiation dose body CT utilizing advanced (model based) iterative reconstruction with a clinical standard radiation dose CT from the same subject. | Baseline (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Y Chen, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2014-H-0188.html